CLINICAL TRIAL: NCT02982772
Title: Biobehavioral Intervention for Smokers Living With HIV (Human Immunodeficiency Virus)
Brief Title: Patch Study - Intervention for HIV Positive Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dr. maria miguez (Other)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor-Investigator, dr. maria miguez, Research Professor, Florida International University
Organization: Florida International University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FloridaIU
Record Dates: First submitted 2016-04-19; First posted 2016-12-05 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Smoking Cessation; HIV
Keywords: Nicotine Replacement; Smoking; HIV
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Combined Modality Therapy; Nicotine; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tailored Combination Therapy (Experimental): Combination of Brief behavioral intervention Plus Nicotine replacement. The test product is a transdermal nicotine patch and Nicotine replacement gums for 12 weeks. The dosage of the test product depends on the amount of cigarettes used.
  Doses will be tailored and adjust as need it
  Interventions: Other: Combination Therapy
- Standard Care Intervention (Active Comparator): Brief behavioral intervention The test product is a transdermal nicotine patch plus regular flavored gums for 10 weeks. The dosage of the test product depends on the amount of cigarettes used.
  Standard Flavored gums will be used as needed for 10 weeks.
  Interventions: Other: Standard Care Intervention

INTERVENTIONS:
Other: Combination Therapy — Brief behavioral intervention
  The test product is a transdermal nicotine patch for 12 weeks. The dosage of the test product depends on the new algorithm (amount, addiction, prior attempts) Nicotine Gums for 12 weeks.
  Other Names: Nicoderm, Nicorette
  Arms: Tailored Combination Therapy
Other: Standard Care Intervention — Brief Behavioral Intervention
  The test product is transdermal Nicotine replacement patch for 10 weeks.The dosage of the test product follows the product guidelines and depends on the amount of cigarettes used.
  Standard Flavored Gums for 10 weeks
  Arms: Standard Care Intervention

SUMMARY:
The overall objective of the transdisciplinary team of Human Immunology Virus (HIV) and Tobacco funded researchers is to test if tailoring nicotine replacement doses to temper these excessive levels will enhance the efficacy of the intervention. To test researchers proposed model 600 people living with HIV (PLWH) ready to quit smokers will be enrolled in a double-blind randomized clinical trial intent-to-treat design, comparing a standard well-validated brief smoking intervention, that following national guidelines + nicotine replacement therapy (NRT), versus the tailored one (brief smoking intervention + personalized doses of nicotine replacement therapy). The primary outcome for this study will be rates of smoking cessation, point prevalence abstinence (prior 7 and prior 30 days), and verified continuous abstinence 3-, 6-, and 12-months post scheduled quit day.

DETAILED DESCRIPTION:
The overall objective of the transdisciplinary team of Human Immunology Virus (HIV) and Tobacco funded researchers is to test if tailoring nicotine replacement doses to temper these excessive levels will enhance the efficacy of the intervention. This will be accomplished by assessing: 1) pre-trial plasma levels, 2) doing genotyping, which to researchers knowledge has not been used in cessation studies among people living with HIV (PLWH), and 3) providing tailored feedback to the participants, based on the assumption that the higher the knowledge and perception of risk, the higher the interest in modifying a risky behavior(s). To test researchers proposed model based in proven smoking prevention and control methods 600 PLWH ready to quit smokers will be enrolled in a double-blind randomized clinical trial intent-to-treat design, comparing a standard well-validated brief smoking intervention, that following national guidelines will consist on brief advice + nicotine replacement therapy, versus the tailored one (brief smoking intervention + personalized doses of nicotine replacement therapy (NRT). The primary outcome for this study will be rates of smoking cessation, point prevalence abstinence (prior 7 and prior 30 days), and verified continuous abstinence 3-, 6-, and 12-months post scheduled quit day. The knowledge gained here has the potential to provide a more complete bio-behavioral model to the intervention field. The proposed study if successful will provide a new tailored, replicable, and manual-based intervention for people living with HIV. It can also provide much need it information in regards to key mediators and moderators of smoking cessation interventions in this vulnerable population. Researchers long term goal is to reduce the burden of one of the most devastating causes of morbi-mortality in researchers time and improve their quality of life. The study could also pave the path to use a similar model to tailor smoking interventions for other populations (e.g., menthol users, older women, adolescents, older adults).

ELIGIBILITY:
Inclusion Criteria:

* HIV infected smokers
* 18 years of age and older
* Fluent in English or Spanish
* Able to consent
* Ready to quit smoking

Exclusion Criteria:

* Psychotic or disabling psychiatric disorders
* Six months post-myocardial infarction or stroke
* Diabetes requiring insulin
* Treatment for vascular problems
* Non-treated hypertension,
* Severe liver or kidney disease
* History of allergies to the nicotine patches
* Severe eczema or psoriasis
* Temporal-mandibular joint disease or dental appliances
* Pregnant women or women that are breastfeeding
* Subjects participating in other interventions/research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2016-05; Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jose Miguez, MD, Principal Investigator — Florida International University; Guillermo Castro, MD, Study Director — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be available only after the study have 2 years of completion. The data to be shared will be de-identified and without data associated with medical records. Access will be provided upon submission of study protocol and if the IRB approves sharing the data.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be available only after two years of study completion
Access Criteria: Requires full disclosure of aims and hypothesis Approval by the center and the IRB committees Signing a limited use agreement

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited with flyers and by referrals.
Pre-assignment Details: 488 participants signed consent forms, a total 11 were excluded (6 did not meet smoking criteria, 3 were not compliant, and 2 had pre-existing medical conditions).
Groups:
- Tailored Combination Therapy: Combination of Brief behavioral intervention Plus Nicotine replacement. The test product is a transdermal nicotine patch and Nicotine replacement gums for 12 weeks. The dosage of the test product depends on the amount of cigarettes used. Doses will be tailored and adjusted as needed.
  Combination Therapy: Brief Behavioral Intervention
  The test product is a transdermal Nicotine patch for 12 weeks. The dosage of the test product depends on the new algorithm (amount, addiction, prior attempts) Nicotine Gums for 12 weeks.
- Standard Care Intervention: Brief behavioral intervention The test product is a transdermal nicotine patch plus regular flavored gums for 10 weeks. The dosage of the test product depends on the amount of cigarettes used.
  Standard Flavored gums will be used as needed for 10 weeks.
  Standard Care Intervention: Brief Behavioral Intervention
  The test product is a transdermal Nicotine replacement patch for 10 weeks.The dosage of the test product follows the product guidelines and depends on the amount of cigarettes used.
  Standard Flavored Gums for 10 weeks
Period: Enrollment
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Started | 245 | 243
Completed | 245 | 243
Not Completed | 0 | 0
Period: Intervention
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Started | 245 | 243
Completed | 226 | 230
Not Completed | 19 | 13
Not completed — Lost to Follow-up | 19 | 13
Period: 1M Follow-Up
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Started | 226 | 230
Completed | 205 | 212
Not Completed | 21 | 18
Not completed — Lost to Follow-up | 21 | 18
Period: 3M Follow-Up
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Started | 205 | 212
Completed | 188 | 201
Not Completed | 17 | 11
Not completed — Lost to Follow-up | 17 | 11
Period: 6M Follow-Up
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Started | 188 | 201
Completed | 177 | 192
Not Completed | 11 | 9
Not completed — Lost to Follow-up | 11 | 9
Period: 12M Follow-Up
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Started | 177 | 192
Completed | 166 | 187
Not Completed | 11 | 5
Not completed — Lost to Follow-up | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored Combination Therapy | Standard Care Intervention | Total
Number analyzed (Participants) | 245 | 243 | 488
Age, Continuous [Mean (Full Range); unit: years] | 50.1 [20 to 69] | 51.1 [21 to 67] | 51.1 [20 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 114 | 212
  Male | 147 | 129 | 276
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic | 33 | 21 | 54
  Race/Ethnicity: Non-Hispanic White | 15 | 20 | 35
  Race/Ethnicity: Non-Hispanic Black | 197 | 202 | 399
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 245 | 243 | 488

OUTCOME MEASURES:

1. Primary Outcome: Rates of Smoking Cessation
Description: verified continuous abstinence (carbon monoxide < 10ppm and cotinine <15 ng/mL).
Time Frame: 3 months
Population: This is the total number of participants in each arm that quit smoking at 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Number analyzed (Participants) | 188 | 201
Participants | 57 | 46

2. Primary Outcome: Rates of Smoking Cessation
Description: verified continuous abstinence (carbon monoxide < 10ppm and cotinine <15 ng/mL).
Time Frame: 6 months
Population: This is the total number of participants in each arm that quit smoking at 6 months. However due to the pandemic we could not verified with biomarkers
Measure: Count of Units; unit: Number of pts that quit
Units Other Than Participants: Number of pts that quit
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Number analyzed (Participants) | 177 | 192
Number analyzed (Number of pts that quit) | 177 | 192
Number of pts that quit | 40 | 28

3. Primary Outcome: Rates of Smoking Cessation
Description: verified continuous abstinence (carbon monoxide < 10ppm and cotinine <15 ng/mL).
Time Frame: 12 months
Population: This is the total number of participants in each arm that quit smoking at 12 months.
Measure: Count of Units; unit: Number of pts that quit
Units Other Than Participants: Number of pts that quit
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Number analyzed (Participants) | 166 | 187
Number analyzed (Number of pts that quit) | 166 | 187
Number of pts that quit | 32 | 28

4. Secondary Outcome: Change in Clinical Outcomes
Description: The investigators will analyze changes in the following parameters since baseline, and will be given one point for each parameter that improves:
  * CD4 (counts and percentage).
  * HIV Viral load (logs).
  * Vital signs (Blood pressure in mm Hg, breaths per minute, beats per minute).
  * Anthropometric measures [Body Mass Index = weight(kilograms) / height(meters2), Waist and hip circumference in inches].
  * In health-related quality of life measured as changes in the total score of Health-Related Quality of Life survey.
  Scale Title: Smoking Cessation Quality of Life (SCQoL) - Physical subscale Minimum 9, maximum 27 (higher scores=worse outcome)
Time Frame: 6 months
Population: Quality of Life change at 6 months.
  Scale Title: Smoking Cessation Quality of Life (SCQoL) - Physical subscale Minimum 9, maximum 27 (higher scores=worse outcome)
Measure: Mean (Standard Deviation); unit: score on a scale/change
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Number analyzed (Participants) | 177 | 192
score on a scale/change | -1.9 (8.8) | 0.38 (7.2)

5. Secondary Outcome: Number of Participants With Verified Continuous Abstinence
Description: Verified continuous abstinence using a breathalyzer carbon monoxide < 10ppm
Time Frame: 3 months
Population: Verified abstinence at 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Number analyzed (Participants) | 188 | 201
Participants | 57 | 46

6. Secondary Outcome: Prevalence of Side Effects-safety
Description: Total number of self reported side effects from Baseline through 6 months.
Time Frame: Baseline-6 months
Population: Total of number of participants in the Tailored & Standard arms.
Measure: Number; unit: side effects
Groups:
- Tailored Combination Therapy: Combination of Brief behavioral intervention Plus Nicotine replacement. The test product is a transdermal nicotine patch and Nicotine replacement gums for 12 weeks. The dosage of the test product depends on the amount of cigarettes used.
  Doses will be tailored and adjust as need it
  Combination Therapy: Brief behavioral intervention
  The test product is a transdermal nicotine patch for 12 weeks. The dosage of the test product depends on the new algorithm (amount, addiction, prior attempts) Nicotine Gums for 12 weeks.
- Standard Care Intervention: Brief behavioral intervention The test product is a transdermal nicotine patch plus regular flavored gums for 10 weeks. The dosage of the test product depends on the amount of cigarettes used.
  Standard Flavored gums will be used as needed for 10 weeks.
  Standard Care Intervention: Brief Behavioral Intervention
  The test product is transdermal Nicotine replacement patch for 10 weeks.The dosage of the test product follows the product guidelines and depends on the amount of cigarettes used.
  Standard Flavored Gums for 10 weeks
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Number analyzed (Participants) | 245 | 243
side effects | 70 | 50

7. Secondary Outcome: Change in Clinical Outcomes
Description: The investigators will analyze changes in the following parameters since baseline, and will be given one point for each parameter that improves:
  * CD4 (counts and percentage).
  * HIV Viral load (logs).
  * Vital signs (Blood pressure in mm Hg, breaths per minute, beats per minute).
  * Anthropometric measures [Body Mass Index = weight(kilograms) / height(meters2), Waist and hip circumference in inches].
  Scale Title: Smoking Cessation Quality of Life (SCQoL) - Physical subscale Minimum 9, maximum 27 (higher scores=worse outcome)
  - In health-related quality of life measured as changes in the total score of Health-Related Quality of Life survey.
Time Frame: 12 months
Population: Quality of Life change at 12 months. Scale Title: Smoking Cessation Quality of Life (SCQoL) - Physical subscale Minimum 9, maximum 27 (higher scores=worse outcome)
Measure: Mean (Standard Deviation); unit: score on a scale/change
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Number analyzed (Participants) | 166 | 187
score on a scale/change | 0.85 (5.9) | 0.82 (5.4)

8. Secondary Outcome: Number of Participants With Verified Continuous Abstinence
Description: verified continuous abstinence using a breathalyzer carbon monoxide < 10ppm
Time Frame: 6 months
Population: Verified abstinence at 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Number analyzed (Participants) | 177 | 192
Participants | 49 | 40

9. Secondary Outcome: Number of Participants With Verified Continuous Abstinence
Description: verified continuous abstinence using a breathalyzer carbon monoxide < 10ppm
Time Frame: 12 months
Population: Verified abstinence at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Number analyzed (Participants) | 166 | 187
Participants | 32 | 28

10. Secondary Outcome: Prevalence of Side Effects-safety
Description: Total number of self reported side effects from 6 through 12 months.
Time Frame: 6 through 12 months
Population: Total of number of participants in the Tailored & Standard arms.
Measure: Number; unit: side effects
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
Number analyzed (Participants) | 245 | 243
side effects | 31 | 33

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Enrollment through the 12 month visit. At each study visit, participants completed a questionnaire regarding side effects.
Arm/Group | Tailored Combination Therapy | Standard Care Intervention
All-Cause Mortality (participants affected / at risk) | 2/245 | 2/243
Serious Adverse Events (participants affected / at risk) | 0/245 | 0/243
Other Adverse Events (participants affected / at risk) | 101/245 | 83/243
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tailored Combination Therapy (N=245) | Standard Care Intervention (N=243)
Jaw Pain (General disorders) | 7 | 6
Dry Mouth (General disorders) | 62 | 49
Skin Rash (Skin and subcutaneous tissue disorders) | 13 | 19
Decrease Appetite (Metabolism and nutrition disorders) | 29 | 22
Headache (Nervous system disorders) | 36 | 44
Dizziness (Nervous system disorders) | 35 | 33
Fatigue (General disorders) | 38 | 39
Sleepiness (General disorders) | 38 | 33
Itching (Skin and subcutaneous tissue disorders) | 31 | 40
Vivid Dreams (Psychiatric disorders) | 1 | 2
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Body Aches (General disorders) | 0 | 3

LIMITATIONS AND CAVEATS:
Please note that verification of quitting was done in all participants before the pandemic. However, during the pandemic the follow up visits were not in person.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT02982772/Prot_002.pdf
  • Statistical Analysis Plan (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT02982772/SAP_001.pdf
  • Informed Consent Form (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT02982772/ICF_003.pdf